CLINICAL TRIAL: NCT06797063
Title: Breastfeeding Education Support Tool
Acronym: BEST4Baby
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); KLE University Jawaharlal Nehru Medical College (Unknown); Benten Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-3092; 1R01HD112492 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Breastfeeding, Exclusive; Infant Development; Infant Growth; Breast Feeding
Keywords: breastfeeding; India; infant feeding; peer counselors
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Participants in the control clusters will continue with local practice for antenatal breastfeeding support and referral to facilities. It is expected that they will receive routine health education recommended by the Indian national health system during the prenatal and postnatal period.
  Interventions: Behavioral: Usual Care
- BEST4Baby (Experimental): BEST4Baby consists of prenatal and post-delivery breastfeeding education and support for mothers provided by community-based peer counselors who are trained in a modified 5-day WHO/UNICEF Breastfeeding Counselling Course and supported by an mHealth application.
  Interventions: Behavioral: BEST4Baby

INTERVENTIONS:
Behavioral: BEST4Baby — BEST4Baby consists of prenatal and post-delivery breastfeeding education and support for mothers provided by community-based peer counselors who are trained in a modified 5-day WHO/UNICEF Breastfeeding Counselling Course and supported by an mHealth application.
  Arms: BEST4Baby
Behavioral: Usual Care — Participants in the control clusters will continue with local practice for antenatal breastfeeding support and referral to facilities. It is expected that they will receive routine health education recommended by the national health system during the prenatal and postnatal period and offered through PHC and community level workers, including ASHAs. ASHAs may visit a woman after delivery to provide lactation support, as needed, with visits ceasing at 42 days post-delivery. Breastfeeding mothers requiring advanced lactation support may be referred to a community subcenter for care with more skilled clinicians.
  Arms: Control

SUMMARY:
The proposed project seeks to evaluate the effectiveness and implementation of the Breastfeeding Education Support Tool for Baby (BEST4Baby) intervention, an mHealth-supported community-based peer counselor breastfeeding intervention for mothers in India. Given that rates of optimal infant feeding practices have remained stagnant over the past two decades in India, and that India is the most populous country and icontributes one-fifth of all global live births, this project could have major global health implications if the intervention is found to improve maternal breastfeeding practices and infant clinical outcomes. The project will also provide evidence needed to adopt BEST4Baby nationally and in other low resource communities.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age,
* pregnant and 20-27 weeks of gestation at study enrollment,
* singleton pregnancy,
* no major antepartum complications,
* living in a research site,
* planning to deliver in the cluster area,
* capable of giving informed consent,
* willing to be visited by a PC and research personnel for up to 12 months post-delivery.

Exclusion Criteria:

comorbidities impacting breastfeeding,

- severe psychological illness that could interfere with consent and study participation. Following a live birth, participants will remain eligible to continue in the study unless the mother or infant experiences: illness or clinical complications warranting prolonged hospitalization, stillbirth, low birth weight (< 2500 g), congenital abnormality, or neonatal death.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study focuses on breastfeeding.
Enrollment: 1152 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
exclusive breastfeeding at 6 months | 6 months
  proportion of infants exclusively breastfed at 6 mo as measured with the infant feeding behavior questionnaire. EBF will be defined as receiving breast milk as the only source of nourishment for the first 6 mo of life, except for oral rehydration solution, vitamins, medicines.
Infant growth velocity | 6 months and 12 months
  mean change in length from birth to 6 months, and birth to 12 months
Infant cognitive development | 12 months
  mean Bayley Scales of Infant and Toddler Development cognitive domain scores at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- KLE Univeristy, Belagavi, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
The survey, anthropometric measurements, and neurodevelopment assessment data will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: All de-identified data will be available upon either publication of related work or completion of the project. The data will be available for at least 10 years after the funding period.